CLINICAL TRIAL: NCT02195245
Title: A New and Innovative Method for CO2 Removal in Anesthetic Circuits: Replacing Chemical Granulate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DMF Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DMF-CLIN-14-01
Record Dates: First submitted 2014-07-11; First posted 2014-07-21 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: End Tidal CO2; CO2 Removal
Keywords: CO2 filter; anesthesia; device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control - Observational (non interventional) data is collected from current state of the art absorber devices.
- memsorb (Experimental): New CO2 filter - data is collected using the new CO2 absorber.
  Interventions: Device: memsorb

INTERVENTIONS:
Device: memsorb
  Arms: memsorb

SUMMARY:
CO2 removal is a mandatory part of modern anesthesia systems. Current chemical absorbers pose problems as the chemical granulate reacts not only with the CO2 but also the anesthetic drugs, producing organ toxic substances. The proposed CO2 absorber provides a solution to the problem of organ-toxin production in anesthetic circuits.

DETAILED DESCRIPTION:
CO2 removal is a mandatory part of modern anesthesia systems. Current chemical absorbers pose problems as the chemical granulate reacts not only with the CO2 but also the anesthetic drugs, producing organ toxic substances. The proposed CO2 absorber provides a solution to the problem of organ-toxin production in anesthetic circuits.

This new absorber can be easily integrated into any anesthesia circuit, and can effectively remove CO2 without reacting with anesthetic drugs, thus eliminating organ-toxic by-products.

It uses advanced membrane technology to separate gas flows within the circuit, separating the expensive anesthetic vapors from the CO2 (the main by-product of metabolism). Anesthetic vapors thus remain in the closed loop circuit, while CO2 is separated and exhausted to the atmosphere, rather than being absorbed through a chemical reaction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Physical Status Class I, II, III (low-medium risk patient)
* English-speaking patients
* Scheduled for elective surgery
* Length of anesthesia ≥ 60 minutes

Exclusion Criteria:

* Pregnant
* American Society of Anesthesiology Physical Status Class IV (high risk patient)
* Patients schedule for emergency surgery
* Known respiratory disease, including COPD and severe asthma
* Have elevated pressure in your brain (intra cranial pressure, ICP)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
End tidal CO2 level | Continuous (5min intervals) over duration of anesthesia. No data collection prior or post anesthesia.
  After completion of the surgery, the digital respiration records are exported from the hospital database.
  End tidal CO2 is assessed as either in range [4.1-5.6]% or out of range <4.1% or >5.6%.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth II HSC, Halifax Infirmary Site, Halifax, Nova Scotia, Canada